Nothing herein is to be disclosed in any way without the prior express written permission of W. L. Gore & Associates, Inc.

# Study of the GORE® EXCLUDER® Endoprosthesis in the treatment Of infra-renal Abdominal Aortic Aneurysms

Protocol number: FPR 12-02

SAP date: 15-NOV-2017

NCT number: NCT02308839

W. L. Gore & Associates, Inc. Medical Products Division

Gore-excluder\_SAP\_V4.0

Sponsor: W.L. GORE

Device : GORE® EXCLUDER®

Protocol Nr: FPR AAA 12-02

# Study of the GORE® EXCLUDER® Endoprosthesis in the treatment of infra-renal Abdominal Aortic Aneurysms (AAA)

Statistical Analysis Plan

| Versions | Date | Documents used / comments |
|---|---|---|
| Version 4.0 | 15/11/2017 | SAP 3.4 |
| | | + SAR comments from WL Gore (by E-mail 19DEC2017) |
| | | + Protocol version 5.1 29FEB2012 |
| Version 3.4 | 13/11/2017 | SAP 3.3 |
| | | + SAR comments from WL Gore (by E-mail 19DEC2017) |
| | | + Protocol version 5.1 29FEB2012 |
| Version 3.3 | 20/12/2017 | SAP 3.2 |
| | | + SAR comments from WL Gore (by E-mail 19DEC2017) |
| | | + Protocol version 5.1 29FEB2012 |
| Version 3.2 | 30/11/2015 | SAP V3.1 |
| | | + SAR comments from WL Gore (26NOV2015) |
| | | + protocol version update |
| | | + Listing 4 title modification |
| | | + Call (30NOV2015) |

### Sponsor:

W.L. Gore & Associés S.A.R.L. 08 place des Vins de France 75012 PARIS France



Gore-excluder\_SAP\_V4.0

Sponsor: W.L. GORE

Device: GORE® EXCLUDER®

Protocol Nr: FPR AAA 12-02

| Versions | Date | Documents used / comments |
|---|---|---|
| Version 3.1 | 26/11/2015 | SAP V3.0 |
| | | + SAR comments from WL Gore (25NOV2015) |
| | | + update of WL Gore address |
| | | + update of signature page |
| | | + update of protocol version |
| | | + update of number of sites involved |
| Version 3.0 | 25/11/2015 | SAP V2.1 |
| | | + SAR comments from WL Gore (19NOV2015) |
| | | + Modification of Table 3, Table 4, Table 5 and Table 28 titles |
| | | + Addition of listing "Implantation main indication" |
| | | + change Listing 5: "Other abnormalities observed" into "Occlusion, stenosis and other abnormalities observed" |
| Version 2.1 | 27/10/2014 | SAP V2.0 |
| | | + Clarification of the SAF population definition |
| | | + Listing 3 title modification |
| Version 2.0 | 13/10/2014 | SAP V1.1 |
| | | + update of AAA following CRF modification |
| Version 1.1 | 26/07/2013 | SAP V1 |
| | | + update of derived criteria calculation section |
| | | + addition of statistical tables and listings |
| Version 1 | 12/04/2013 | Protocol Number FPR AAA 12-02 (Version 5.1) |



Gore-excluder\_SAP\_V4.0.doc
Sponsor: W.L. GORE

Device : GORE® EXCLUDER®

Protocol Nr: FPR AAA 12-02

# SIGNATURE PAGE

# STUDY OF THE GORE® EXCLUDER® ENDOPROSTHESIS IN THE TREATMENT OF INFRA-RENAL ABDOMINAL AORTIC ANEURYSMS (AAA)

### Version 4.0

# W.L. GORE & ASSOCIÉS S.A.R.L.

| Name | Position | Date | Signature |
|------------------|--------------------------|-------------|-----------|
| Abe Letter | Clinical Biostatistician | 15-NOV-2018 | Ohe Sth |
| Alexandre Figard | Clinical Study Manager | 19-NOV-2018 | AM |
| | | | N. |






# **TABLE OF CONTENTS**

STATISTICAL ANALYSIS PLAN

| 1. | Over | view | | 6 |
|---|---|---|---|---|
| | 1.1. | Study ( | Objective | 6 |
| | 1.2. | Study I | Design | 6 |
| | 1.3. | _ | Plan | |
| | | 1.3.1. | Sample Size | |
| | | 1.3.2. | Patient's Follow-up | 6 |
| | | 1.3.3. | Study Device | 6 |
| | | 1.3.4. | Study Assessments | 7 |
| 2. | Stati | stical m | nethods | 7 |
| | 2.1. | Genera | al Statistical Considerations | 7 |
| | | 2.1.1. | Time Points Definition | |
| | | 2.1.2. | Derived Criteria Calculation | |
| | | 2.1.3. | Handling Missing Data | |
| | | 2.1.4. | Descriptive Statistics in Summary Tables | |
| | | 2.1.5. | Inferential Analysis | |
| | | 2.1.6. | Data Listings | |
| | 2.2. | • | e size calculation | |
| | 2.3. | Analys | is Sets | |
| | | 2.3.1. | Definition of patient populations | 9 |
| | 2.4. | Statistic | cal Analyses | |
| | | 2.4.1. | Patient Disposition | |
| | | 2.4.2. | Patient Characteristics | |
| | | 2.4.3. | Endpoints Analyses | |
| | | 2.4.4. | Safety analysis | 11 |
| 3. | Stati | stical S | oftware | 11 |
| 4. | Layo | ut of th | ne statistical tables | 12 |
| | 4.1. | Quantit | tative variables | 12 |
| | | 4.1.1. | ·· | |
| | | 4.1.2. | By group (Type 2) | 12 |
| | 4.2. | Qualita | ative variables | 12 |
| | | 4.2.1. | 777'd ( | |
| | | | Without group (Type 3) | |
| | | 4.2.1. | By group (Type 4) | 13 |
| | | 4.2.2. | By group (Type 4)<br>Conditional variables (Type 5) | 13 |
| | 4.3. | 4.2.2. | By group (Type 4) Conditional variables (Type 5) type of tables | 13<br>13 |
| | 4.3. | 4.2.2.<br>Other t<br>4.3.1. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) | 13<br>13<br>13 |
| | 4.3. | 4.2.2.<br>Other t<br>4.3.1.<br>4.3.2. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) | 13<br>13<br>13<br>13 |
| | 4.3. | 4.2.2.<br>Other t<br>4.3.1. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) | 13<br>13<br>13<br>13 |
| 5. | | 4.2.2.<br>Other t<br>4.3.1.<br>4.3.2.<br>4.3.3. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) | |
| 5. | | 4.2.2.<br>Other t<br>4.3.1.<br>4.3.2.<br>4.3.3.<br>e of con | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) | |
| 5. | Tabl | 4.2.2.<br>Other t<br>4.3.1.<br>4.3.2.<br>4.3.3.<br>e of con | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) | |
| 5. | Tabl | 4.2.2.<br>Other t<br>4.3.1.<br>4.3.2.<br>4.3.3.<br>e of con<br>Tables. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) Itents Patient Disposition Patient Characteristics | |
| 5. | Tabl | 4.2.2. Other t 4.3.1. 4.3.2. 4.3.3. e of con Tables. 5.1.1. 5.1.1. 5.1.2. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) Atents Patient Disposition Patient Characteristics Endpoint analysis | |
| 5. | Tabl | 4.2.2. Other ty 4.3.1. 4.3.2. 4.3.3. e of con Tables. 5.1.1. 5.1.2. 5.1.3. | By group (Type 4) Conditional variables (Type 5) ype of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) ntents Patient Disposition Patient Characteristics Endpoint analysis Safety Analysis | |
| 5. | Tabl | 4.2.2. Other ty 4.3.1. 4.3.2. 4.3.3. e of con Tables. 5.1.1. 5.1.2. 5.1.3. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) Tents Patient Disposition Patient Characteristics Endpoint analysis Safety Analysis | |
| 5. | <b>Tabl</b> 5.1. | 4.2.2. Other t 4.3.1. 4.3.2. 4.3.3. e of con Tables. 5.1.1. 5.1.2. 5.1.3. Listing. 5.2.1. | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) Tents Patient Disposition Patient Characteristics Endpoint analysis Safety Analysis Safety Analysis Patient Disposition | |
| 5. | <b>Tabl</b> 5.1. | 4.2.2. Other t 4.3.1. 4.3.2. 4.3.3. e of con Tables. 5.1.1. 5.1.2. 5.1.3. Listing: | By group (Type 4) Conditional variables (Type 5) type of tables Flowchart (Type 6) Adverse Events (Type 9) Survival curve (Type 10) Tents Patient Disposition Patient Characteristics Endpoint analysis Safety Analysis | |

# List of abbreviations and definition of terms

| AAA | Abdominal Aortic Aneurysms |
|------|------------------------------------------|
| AE | Adverse Event |
| FUP | Follow-up |
| ICU | Intensive Care Unit |
| ITT | Intent-To-Treat population |
| LPP | List of products |
| LPPR | List of products and refundable services |
| SAF | Safety population |
| SAP | Statistical Analysis Plan |



### OVERVIEW

This statistical analysis plan (SAP) describes the planned statistical analyses of the data collected in the course of the Register Gore® Excluder® AAA France.

This SAP provides additional details concerning the statistical analyses outlined in the protocol (version dated 29FEB2012). The purpose of the SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches to the analysis of study data.

### 1.1. Study Objective

The objective of this study is to assess the usefulness of the technique by documenting overall mortality, complications (endoleak, migration), the rate of surgical conversion, the evolution and rupture of the aneurysm, in the long term, that is, 5 years, on a cohort of patients representative of the population treated in real life conditions.

### 1.2. Study Design

The study is a observational, prospective and multicentric register of the GORE® EXCLUDER® AAA Endoprosthesis used to treat infrarenal abdominal aortic aneurysms in which 180 patients are enrolled from 29 sites and followed during 5 years minimum.

### 1.3. Study Plan

### 1.3.1. Sample Size

A total of 180 patients are enrolled in this study,

### 1.3.2. Patient's Follow-up

8 visits are scheduled:

- Visit 1 : Baseline
- Visit 2 : Procedure
- Visit 3 : Discharge
- Visit 4 : Post operatory (or in the month following the surgery)
- Visit 5: 6 months Follow-up
- Visit 6: 1 year Follow-up
- Visit 7: 2 years Follow-up
- Visit 8: 3 years Follow-up
- Visit 9: 4 years Follow-up
- Visit 10: 5 years Follow-up

### 1.3.3. Study Device

The studied device is the GORE® EXCLUDER® Endoprosthesis and any evolution registered on LPP.

### FPR AAA 12-02


### STATISTICAL ANALYSIS PLAN

### 1.3.4. Study Assessments

The following flowchart applies to the study:

| | Post operatory<br>follow-up<br>(D1 à D30) | Follow-up at 6<br>months | Follow-up at 1, 2, 3, 4 and 5 years | Intermediate<br>follow-up*** |
|---|---|---|---|---|
| Clinic exam | x | x | x | x |
| Abdominal X-ray without preparation under 3 angles (face, profile and 3/4) | X1 | X* | X* | X* |
| Tomography with contrast product | х | x | x | х |
| MRI | X* | X* | X* | X* |
| Vascular echo-doppler | X** | X** | X** | X** |

<sup>\*</sup> if tomography with contrast product cannot be performed

### 2. STATISTICAL METHODS

### 2.1. General Statistical Considerations

### 2.1.1. Time Points Definition

Baseline data is defined as the last available observation recorded before the first study device exposition for the patient.

Visit(n) data is defined as the last available observation on or before the Visit(n) time point following the first study device exposition for the patient.

Endpoint data is defined as the last follow-up at 5 years or, if the data is missing, as the last available observation recorded for the patient.

If the hospital discharge visit did not occur before the post-operatory follow-up, it will be considered as an unscheduled visit.

### 2.1.2. Derived Criteria Calculation

- · Age classes will be the following:
  - o Age < 80 years
  - o Age ≥ 80 years
- · Body Mass Index will be calculated as :
  - $BMI = weight (kg) / (height (m))^2$
- Duration between two dates i and j will be calculated as:
  - Duration i, j = Date j Date i +1
- If no clinical exam is done at a particular visit, the visit date will be the last imaging exam date reported for this visit.
- · Total study duration will be calculated as:
  - Total study duration = study exit date procedure date +1
  - If the procedure date is not available, the baseline will be used instead.

<sup>\*\*</sup> If MRI cannot be performed

<sup>\*\*\*</sup> Intermediate follow up are realized only if leak, deterioration of endoprosthesis or evolution of aneurysms are noticed in the last follow up. The follow-up needs to be done within 3 months after the exam which noticed the anomaly.

<sup>&</sup>lt;sup>(1)</sup> Radiography in postoperative follow-up will not be necessary in case of 3D reconstruction performed during tomography.

FPR AAA 12-02


- · Study follow-up duration will be calculated as:
  - Study follow-up duration = last FUP date available procedure date +1
  - If the procedure date is not available, the baseline will be used instead.
- · Surgical risk for patient (AFSSAPS' criteria):

A patient is considered as "at high risk" (surgical risk = High instead of Normal) if at least one of the following criteria is met:

- o Age ≥ 80 years
- Coronary artery disease (history of myocardial infarction or angina) with positive functional testing and coronary lesions for which revascularization is impossible or not indicated
- Cardiac failure with patent clinical manifestations
- Inoperable aortic stenosis
- LVEF < 40 %</li>
- o Chronic respiratory failure objectified by one of the following criteria
  - FEV < 1.2 l/sec</li>
  - VC < 50% of the predicted value according to age, sex and weight</li>
  - Arterial blood gases in the absence of oxygen: PaCO<sup>2</sup> > 45 mm Hg or PaO<sup>2</sup> < 60 mm Hg</li>
  - Home Oxygen Therapy
- Renal failure, if serum creatinine > 200 μmol / L before injection of contrast medium
- Hostile abdomen, including the presence of ascites or other signs of portal hypertension
- If more than one imaging technique are used to measure the maximum AAA diameter, and all the
  measures are not the same, the maximum AAA diameter will be the one measured by the more
  precise technique based on the following:

CT with contrast > MR with contrast > CT without contrast > MR without contrast > Echo Doppler

More precise

Less precise

- . The maximum aneurysm diameter classes will be the following:
  - o "Small": maximal AAA diameter less than 5 cm
  - "Average": maximal AAA diameter between 5 and 7 cm
  - o "Large": maximal AAA diameter more than 7 cm
- The diameter increase will be analyzed as follows:

If the diameter observed is at least 5 mm greater than the largest aneurysm diameter (observed at the first post-op control) then there is a diameter increase.

- The migration will be analyzed as follows:
  - Distal migration is defined as a distal movement strictly greater than 10 mm since the first post-op control.
  - A proximal migration is defined by a proximal movement either strictly greater than 10 mm or which covers one of the renal arteries since the first post-op control.

If at least one of the two migrations is observed then migration = "Yes"

· Endoleak will be analyzed as follows:

If an endoleak (I, II or III) appears during follow-up then Endoleak = "Yes"

### 2.1.3. Handling Missing Data

No replacement of missing data is planned.

In case of missing data, the patient will be considered as censured at his/her last available observation in survival analyses.

In case of partially missing death dates (day of death missing) confirmed as unknown by the site, the first day of the month will be imputed. If the death occurs in the same month as last follow-up then the later day of the two will be imputed.

### FPR AAA 12-02


### STATISTICAL ANALYSIS PLAN

### 2.1.4. Descriptive Statistics in Summary Tables

- Continuous variables will be summarized using standard quantitative statistics: number of nonmissing observations, mean, standard deviation, median, quartiles and range (minimum and maximum observed values). The number of missing observations will also be specified.
- Categorical variables will be summarized using classical frequency statistics: number of non-missing observations and percentages by categories. Percentages will be calculated on the number of non-missing observations, and will be displayed using one decimal. The number of missing observations will also be specified.

### 2.1.5. Inferential Analysis

No inferential analysis is planned for the first analysis part of this study.

### 2.1.6. Data Listings

Patient data listings will be selected to be supportive of summary statistical tables, including derived/calculated data from statistical process. These key data listings will be performed on selected analysis sets according to the focus of the listings and will be sorted by patient number or visit.



### 2.3. Analysis Sets

### 2.3.1. Definition of patient populations

2 populations will be defined:

- The Safety (SAF) population will include all patients enrolled in the study and who have signed their informed consent or accept the use of their data.
- The Intent-to-Treat (ITT) population will include all safety patients who underwent surgery (i.e. who
  used at least one GORE® EXCLUDER® AAA Endoprosthesis).

### 2.4. Statistical Analyses

### 2.4.1. Patient Disposition

All the following tables will be presented on SAF population instead otherwise described.

- The number of patients included/non included will be presented by sites.
- A study flowchart table will be presented on SAF and ITT populations.
- The number of patients withdrawn will be presented by reason of interruption and a list of these reasons will be provided.
- Study duration:
  - The total study duration (between procedure and study exit) will be presented globally.
  - The study follow-up duration (between procedure and the last available follow-up) will also be presented in intermediary report(s).

FPR AAA 12-02


· All deviations reported by the investigators will be listed.

### 2.4.2. Patient Characteristics

Descriptive statistics will be used to draw up a recapitulation of ITT patients characteristics at baseline and procedure.

### 2.4.2.1. Baseline

- Demographics
- Medical condition
- Surgical Risk
- · Aneurysm characteristics

### 2.4.2.2. Procedure

- Implantation main indication (a listing will also be presented).
- Implantation parameters (all patients not implanted with GORE® EXCLUDER® AAA Endoprosthesis bifurcated will be listed)
- Procedure evaluation and results (a listing of all associated surgical/endovascular procedures details and a listing of all other abnormalities observed will be presented)
- GORE® EXCLUDER® AAA Endoprosthesis details (listing)
- Discharge: Stay in ICU

### 2.4.3. Endpoints Analyses

The endpoint analyses will be performed on the ITT population.

Primary analysis consists to study the 5-year mortality of patients who received the endoprosthesis. Secondary analyses consist to study the other safety parameters on patients who received the endoprosthesis.

The dates to be used for the "aneurysm diameter evolution" survival analysis will be the date of the imaging exam on which it has been reported. If it is missing, the corresponding "clinical exam" date will be used instead.

The same will be done for the "endoleak complication" and "device migration" survival analyses.

### 2.4.3.1. Primary Analysis

The 5-year mortality survival curve will be described according to the Kaplan-Meier method. The associated Kaplan-Meier estimators will be calculated. Only events occurring up to 5 years (1826 days) of follow-up will be analyzed for mortality survival curve.

### 2.4.3.2. Secondary Analyses

The surgical conversion rate during procedure and the corresponding 95% confidence interval will be provided.

The following parameters will be presented using the Kaplan-Meier survival curves:

- · Mortality related to the aneurysm
- · Aneurysm diameter evolution
- Endoleak complication, for each type (I, II and III)
- Device migration overall and by type (distal, proximal)
- Re-intervention

For the parameters "Aneurysm diameter evolution", "Endoleak complication" and "Device migration", the date to be used for the survival analysis is the date of the first visit where the parameter is reported. Only events occurring up to 5 years (1826 days) of follow-up will be analyzed for these survival curves.

# 

# 3. STATISTICAL SOFTWARE

All statistical outputs (summary tables and data listings) will be generated using SAS® version 9.4 or later.




### 4. LAYOUT OF THE STATISTICAL TABLES

### 4.1. Quantitative variables

# 4.1.1. Without group (Type 1)

| | N | Missing | Mean | S.D. | Median | Min,Max | Q1-Q3 |
|----------|----|---------|------|------|--------|-----------|-------------|
| Variable | XX | XX | XX,X | XX,X | XX,X | XX,X,XX,X | XX,X - XX,X |

# 4.1.2. By group (Type 2)

| | Group | N | Missing | Mean | S.D. | Median | Min,Max | Q1-Q3 |
|---|---|---|---|---|---|---|---|---|
| Variable | Group 1 | XX | XX | XX,Z | XX,Z | XX,Z | XX,Z, XX,Z | XX,Z - XX,Z |
| | Group 2 | XX | XX | XX,Z | XX,Z | XX,Z | XX,Z, XX,Z | XX,Z - XX,Z |
| | Total* | XX | XX | XX,Z | XX,Z | XX,Z | XX,Z , XX,Z | XX,Z - XX,Z |

### 4.2. Qualitative variables

# 4.2.1. Without group (Type 3)

| | | POP<br>(N=XX) |
|----------|-----------------|---------------|
| Variable | N | XX |
| | Mod 1 | XX (XX.X%) |
| | IC 95% (Mod 1)* | [XX.X; XX.X] |
| | Mod n | XX (XX.X%) |
| | IC 95% (Mod n)* | [XX.X; XX.X] |
| | Missing | XX |

<sup>\*</sup> if needed


# 4.2.1. By group (Type 4)

| | | | Group | |
|---|---|---|---|---|
| | | Group 1<br>(N=XX) | Group 2<br>(N=XX) | Total*<br>(N=XX) |
| Variable | N | XX | XX | XX |
| | Mod 1 | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | IC 95% (Mod 1)* | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| | Mod n | XX (XX.X %) | XX (XX.X %) | XX (XX.X %) |
| | IC 95% (Mod n)* | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| | Missing* | XX | XX | XX |

<sup>\*</sup> if needed

# 4.2.2. Conditional variables (Type 5)

| ∨ariable<br>/ Conditional variable | Population*<br>(N=XX) | Group 1*<br>(N=XX) | <br>Group n*<br>(N=XX) |
|---|---|---|---|
| Mod 1 | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |
| Conditional Mod 1 | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |
| | | | <br> |
| Conditional Mod n | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |
| | | | <br> |
| Mod n | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |
| Conditional Mod 1 | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |
| | | | <br> |
| Conditional Mod n | XX (XX.X %) | XX (XX.X %) | <br>XX (XX.X %) |

<sup>\*</sup> if needed

# 4.3. Other type of tables

# 4.3.1. Flowchart (Type 6)

| Populations / Reasons | SAF population | ITT Population |
|-----------------------|----------------|----------------|
| Baseline | XX (XX.X %) | XX (XX.X %) |
| Study exit reason 1* | XX (XX.X %) | XX (XX.X %) |
| Study exit reason 2* | XX (XX.X %) | XX (XX.X %) |
| 5 Year FUP* | XX (XX.X %) | XX (XX.X %) |

<sup>\*</sup> if any



### Page 14/17

# 4.3.2. Adverse Events (Type 9)

| | POP<br>(N=XX) | | |
|----------------|---------------|----------|----------|
| Adverse events | NAE<br>(1) | n<br>(2) | %<br>(3) |
| AE type 1 | XX | XX | XX.X |
| AE type 2 | XX | XX | XX.X |
| | XX | XX | XX.X |
| AE type n | XX | XX | XX.X |

STATISTICAL ANALYSIS PLAN

- (1): Number of adverse events
- (2): Number of patients
- (3): (n / N)\*100 (N: number of patients)

## 4.3.3. Survival curve (Type 10)



### Summary table

| | Mod 1<br>(n=X) | <br>Mod n*<br>(n=X) |
|----------------------------------|----------------|---------------------|
| Nb of patients | х | <br>X |
| Nb of patients with an event | X (XX.XX%) | <br>X (XX.XX%) |
| Nb of patients without an event | X (XX.XX%) | <br>X (XX.XX%) |
| Survival rate | XX % | <br>XX % |
| Progression-Free survival (days) | | |
| Median | XX | <br>XX |
| (95% CI) | (XX, XX) | <br>(XX, XX) |
| 25th-75th percentile | XX.X – XX.x | <br>XX.X – XX.x |
| Range | X - X | <br>X - X |

<sup>\*</sup> If any



### TABLE OF CONTENTS

### 5.1. Tables

### 5.1.1. Patient Disposition

Table 1 : Patients status by sites (Type 4)

Table 2: Study flowchart (Type 6)

Table 3: Withdrawals and study exit reasons (Type 3)

Table 4: Study durations (days) (Type 1)

### 5.1.1. Patient Characteristics

### 5.1.1.1. Baseline

Table 5 : Age at surgery (years) (Type 1)

Table 6: Age classes at surgery (Type 3)

Table 7 : Gender (Type 3)

Table 8: Weight (kg) (Type 1)

Table 9: Height (cm) (Type 1)

Table 10 : BMI (Type 1)

Table 11 : Medical history (Type 3)

Table 12: ASA classification (Type 3)

Table 13: Surgical risk (Type 3)

Table 14: Maximal aneurysm diameter (mm) (Type 1)

Table 15: Maximal aneurysm diameter classes (Type 3)

Table 16: Angle between proximal aortic neck and main axis of the AAA (degrees) (Type 1)

Table 17: Proximal neck length (mm) (Type 1)

Table 18: Proximal neck diameter (mm) (Type 1)

Table 19: Proximal aortic neck characteristics (Type 3)

### 5.1.1.2. Procedure

Table 20: Implantation main indication (Type 3)

Table 21: Duration of procedure (minutes) (Type 1)

Table 22: GORE® EXCLUDER® AAA Endoprosthesis bifurcated (Type 3)

Table 23 : Access type (Type 3)

Table 24: Type of anesthesia used (Type 3)

Table 25: Volume of contrast medium (ml) (Type 1)

Table 26: Time under fluoroscopy (minutes) (Type 1)

Table 27: Procedure outcome and failure details (Type 3)

Table 28: Related surgical/endovascular procedures (Type 3)

Table 29 : Surgical complications (Type 3)

Table 30 : Abnormalities observed (Type 5)

Table 31 : Endoleak (Type 5)

Table 32 : Stay in Intensive Care Unit (hours) (Type 1)

FPR AAA 12-02


### 5.1.2. Endpoint analysis

### 5.1.2.1. Primary Analysis

Table 33: Mortality survival analysis (Type 10)

5.1.2.2. Secondary Analysis

- Table 34 : Surgical conversion rate (Type 3)
- Table 35: Mortality related to aneurysm survival analysis (Type 10)
- Table 36: Diameter increase survival analysis (Type 10)
- Table 37: Endoleak survival analysis overall (Type 10)
- Table 38 : Endoleak survival analysis type I (Type 10)
- Table 39 : Endoleak survival analysis type II (Type 10)
- Table 40 : Endoleak survival analysis type III (Type 10)
- Table 41: Migration survival analysis overall (Type 10)
- Table 42: Migration survival analysis distal (Type 10)
- Table 43: Migration survival analysis proximal (Type 10)
- Table 44: Re-intervention survival analysis (Type 10)



### 5.2. Listings

### 5.2.1. Patient Disposition

Listing 1: Withdrawals

Listing 2: Deviations as reported by investigators

### FPR AAA 12-02


### 5.2.2. Patient Characteristics

### 5.2.2.1. Procedure

- Listing 3: Implantation main indication
- Listing 4: Patient not implanted with GORE® EXCLUDER® AAA Endoprosthesis bifurcated

STATISTICAL ANALYSIS PLAN

- Listing 5: Associated surgical/endovascular procedures
- Listing 6: GORE® EXCLUDER® AAA Endoprosthesis details